CLINICAL TRIAL: NCT05056454
Title: Perinatal Mood Tracking and Treatment
Brief Title: New Moms Mood Tracking & Wellbeing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Michelle Craske, Distinguished Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20-001924
Record Dates: First submitted 2021-07-12; First posted 2021-09-24 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Depression; Perinatal Depression; Anxiety; Pregnancy Related
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Perinatal Psychiatric Care (Other): This treatment condition is modelled after the psychiatry-delivered treatment usually provided at the Maternal Outpatient Mental Health Services (MOMS) Clinic associated with the UCLA Westwood OB-GYN Clinic and Department of Psychiatry.
  Interventions: Other: Perinatal Psychiatric Care
- Screening and Treatment of Anxiety and Depression (STAND) (Experimental): This treatment condition provides access to a system of care, in which type of treatment is allocated based on presenting symptomatology. Participants will learn their allocation from study staff or participants will create a secure account through STAND to learn about their allocation through the STAND online dashboard. Through their STAND online dashboard, they could also have access to their CAT-MH results over time from the start of treatment.
  Interventions: Behavioral: Online therapy with coaching within STAND; Behavioral: Clinical care within STAND

INTERVENTIONS:
Behavioral: Online therapy with coaching within STAND — Participants with moderate depressive symptoms on the CAT-MH (and no current suicidality) will meet with a trained coach, and receive access to online course materials from one of 2 lesson platforms - ThisWayUp's MUMentum course or UCLA DGC's ParentMood course. The efficacy of each online course will be compared for equivalency.
  Participants are encouraged to practice their lesson homework for at least one week before meeting with their coach and starting the next lesson.
  Arms: Screening and Treatment of Anxiety and Depression (STAND)
Behavioral: Clinical care within STAND — Participants with severe depressive symptoms or significant suicidality on the CAT-MH will be allocated to access clinical care, which entails weekly psychotherapy sessions and psychiatric care, when needed or appropriate. While clinical care will be available for the entire 6-month duration of the treatment component of the study, participants will be informed that on average therapy is completed within 13 sessions. The schedule of psychiatric care will be determined by the provider.
  Arms: Screening and Treatment of Anxiety and Depression (STAND)
Other: Perinatal Psychiatric Care — Perinatal psychiatric care involves medication management and supportive therapy for up to six months, with referrals to relevant community resources by the final visit.
  Arms: Perinatal Psychiatric Care

SUMMARY:
New moms can be at risk for perinatal depression (PND). The New Moms Mood Tracking and Wellbeing study is investigating mood changes, risk factors for depression and anxiety and treatment response around the time of delivery. Participants will be asked to complete three sets of online surveys between week 28 gestation and week 20 after delivery, in addition to downloading an app to collect data using their smartphone sensors and brief symptom surveys every other week. Women with elevated symptoms will be eligible to participate in a treatment study. Women who are eligible for the treatment study will be randomized to one of two conditions - Perinatal Psychiatric Care or Screening and Treatment for Anxiety and Depression (STAND). In Perinatal Psychiatric Care, participants will receive appointments with psychiatry clinicians for medication management and supportive therapy. In STAND, participants will be allocated to Online therapy with Coaching or Clinical Care, which includes both psychotherapy and psychiatry appointments. Treatment can last up to 6 months and there will be treatment related assessments for the duration of the 6 months, in addition to brief symptom surveys on a regular basis. Therefore, participation can last between 24 and 52 weeks, as both time of delivery and treatment enrollment timepoint cannot be scheduled in advance.

ELIGIBILITY:
Inclusion Criteria:

* Women who are between week 28 of their pregnancy and 6 months postpartum and are receiving care at a UCLA OB-GYN clinic
* Fluent in English
* Current endorsement of moderate or higher depression on the Edinburgh Postnatal Depression Scale (EPDS, => 11 sum score), administered by the treating OB-GYN physician or study staff
* Not currently in individual treatment for a behavioral or emotional problem (e.g., anxiety, depression)
* Willingness to follow study procedures
* Willingness to participate in treatment through the study and follow all study procedures, including provide HIPAA Authorization for research
* Has access to the internet via mobile or desktop device

Exclusion Criteria:

* Are currently receiving treatment by a therapist or a psychiatrist
* Unstable suicidality (e.g., 2 or more suicide attempts or self-injurious behaviors resulting in hospitalization in the last 6 months, combined with high ratings on self-reported negative urgency)
* Current substance use disorder that interferes with treatment: specifically, patients meeting diagnostic criteria for Substance Use Disorder (SUD) will be eligible for inclusion only if they are able to attend sessions while not under the influence of that substance, with the exception of individuals abusing opiates or freebase cocaine, who will be excluded
* Principal diagnosis of psychosis unrelated to depression (unipolar or bipolar)
* Neurological conditions
* Severe uncontrolled medical conditions (e.g., anorexia nervosa, cardiac conditions requiring continuous monitoring)
* Cognitive impairment (e.g., developmental disability, dementia)

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Computerized Adaptive Testing - Mental Health (CAT-MH) Scores every two weeks until Week 26 | Week 2-26
  Evaluation of degree of change in depression score throughout and after defined treatment periods as measured by the CAT-MH scores.
  The CAT-MH uses item response theory (IRT) to select a subset of items from a pool of approximately 1000 questions to target the respondent's impairment level. It consists of five modules, which screen for a diagnosis of Major Depressive Disorder, depressive symptoms, anxiety symptoms, mania, and suicidal ideation.

SECONDARY OUTCOMES:
Edinburgh Postnatal Depression Scale (EPDS-9) | Post-treatment and week 26
  Evaluation of degree of change in depression score after defined treatment periods as measured by the Edinburgh Postnatal Depression Scale (EPDS-9) scores.
  The Edinburgh Postnatal Depression Scale (EPDS-9) is a 9-item version of the Edinburgh Postnatal Depression Scale (EPDS-10), which omits the 10th item ("The thought of harming myself has occurred to me") of the original 10-item Edinburgh Postnatal Depression Scale.
  The 9 items are summed into a single score ranging from 0 (depression not likely) to 27 (probable depression).

OTHER OUTCOMES:
Sheehan Disability Scale (SDS) | Week 26
  The Sheehan Disability Scale (SDS) is a self-report measure which assesses functional impairment in three inter-related domains; work/school, social and family life.The three items asking about work, social life, and family life are rated on a scale of 0-10 where:
  0 = Not at all 1-3 = Mildly 4-6 = Moderately 7-9 = Markedly 10 = Extremely
  The 3 items can also be summed into a single dimensional measure of global functional impairment that ranges from 0 (unimpaired) to 30 (highly impaired).

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Los Angeles (UCLA), Los Angeles, California, United States

REFERENCES:
- [Derived] Wolitzky-Taylor K, Richards MC, Welborn A, McDonald V, Arnaudova I, Fears S, O'Mahen H, Newby JM, Millard M, Metts AV, Stein A, Freimer N, Craske MG. Study protocol: perinatal mood treatment study. Trials. 2024 Aug 6;25(1):525. doi: 10.1186/s13063-024-08086-w. PMID 39107820